CLINICAL TRIAL: NCT04972981
Title: A Phase 1, Open-Label, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ADCT-901 as Monotherapy in Patients With Selected Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ADCT-901 in Participants With Selected Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-901-101; 2021-002292-19 (EudraCT Number)
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumors
Keywords: Advanced Solid Tumors; ADCT-901

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): In Part 1 (dose escalation) participants with selected advanced solid tumors will receive escalating doses of ADCT-901 as monotherapy. Participants can receive ADCT-901 until disease progression, adverse event (AE), or other discontinuation criteria, whichever occurs first.
  Interventions: Drug: ADCT-901
- Part 2: Dose Expansion (Experimental): In Part 2 (dose expansion), participants will receive ADCT-901 monotherapy at the dose identified as the RP2D/MTD in Part 1 (dose escalation).
  Participants will be split into two groups:
  Group 1: An indication for which ADCT-901 showed in Part 1 to have preliminary activity.
  Group 2: A group of participants with Part 1 indications, except for the one selected in Group 1 of Part 2. No more than 30% of participants with the same indication are allowed in this basket group.
  Participants can receive ADCT-901 until disease progression, AE, or other discontinuation criteria, whichever occurs first.
  Interventions: Drug: ADCT-901

INTERVENTIONS:
Drug: ADCT-901 — Intravenous infusion

SUMMARY:
The primary objectives of this study are to identify the recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD), and to characterize the safety and the tolerability of ADCT-901.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologic diagnosis of selected solid tumor malignancy that is locally advanced or metastatic at time of Screening: cholangiocarcinoma, ovarian/fallopian tube cancers, prostate cancer, renal cell carcinoma, and triple negative breast cancer (TNBC).

   Note: Histologic variants of prostate cancer, including neuroendocrine features and small cell carcinoma of the prostate are permitted.
2. Participants who are refractory to or intolerant to existing therapy(ies) known to provide clinical benefit for their condition per Investigator judgment.
3. Participants with measurable disease as determined by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1:

Note 1: Lytic bone lesions or mixed lytic-blastic lesions, with identifiable soft tissue components, that can be evaluated by cross sectional imaging techniques such as computed tomography (CT) or magnetic resonance imaging (MRI) can be considered as measurable lesions only if the soft tissue component meets the definition of measurability per RECIST v1.1.

Note 2: Prostate cancer participants without measurable lesions will be accepted, with evidence of bone metastatic disease on radiographic examination, whether from bone scan or other imaging modality, and prostate specific antigen (PSA) ≥2.0 ng/mL.

Exclusion Criteria:

1. History of active infection (requiring intravenous [IV] antibiotics, IV antiviral or IV antifungal treatment within 4 weeks of cycle 1, day 1 [C1D1]).
2. Symptomatic central nervous system (CNS) metastases or evidence of leptomeningeal disease (brain MRI or previously documented cerebrospinal fluid cytology). Previously treated asymptomatic CNS metastases are permitted provided that the last treatment (systemic anticancer therapy and/or local radiotherapy) was completed ≥4 weeks prior to C1D1 except usage of low dose of steroids on a taper (i.e., up to 10 mg prednisone or equivalent on Day 1 and consecutive days is permissible if being tapered down). Participants with discrete dural metastases are eligible.
3. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or any serosal effusion that is either requiring drainage or associated with shortness of breath).
4. Active diarrhea ≥ Common Terminology Criteria for Adverse Events (CTCAE) Grade 2 or a medical condition associated with chronic diarrhea (such as irritable bowel syndrome, inflammatory bowel disease).
5. Active or clinically significant ocular surface disease at baseline. An ocular evaluation is to be confirmed by an ophthalmologist at screening. Participants with any prior episode of cicatricial conjunctivitis (as evaluated by the investigator) are ineligible.

   Note: Mild dry eye syndrome or blepharitis managed with artificial tear drops, without injection or epithelial changes, are not exclusionary.
6. Use of any other experimental medication within 14 days prior to start of study drug (C1D1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) | Up to approximately 2.5 years
  Adverse events (AEs) and serious adverse events (SAEs) were defined as any untoward medical occurrence in participants whether or not considered related to the investigational medicinal product. Any clinically significant changes in vital signs, laboratory values, 12-lead electrocardiogram (ECG) and Eastern Cooperative Oncology Group (ECOG) performance status results will be recorded as AEs and SAEs.
Number of Participants Who Experience a Dose Limiting Toxicity (DLT) During the Dose-Escalation Phase | Day 1 to Day 21
Number of Participants Who Experience a Dose Interruption | Up to approximately 2.5 years
Number of Participants Who Experience a Dose Reduction | Up to approximately 2.5 years

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 2.5 years
Duration of Response (DOR) | Up to approximately 2.5 years
Progression-Free Survival (PFS) | Up to approximately 2.5 years
Overall Survival (OS) | Up to approximately 2.5 years
Maximum Concentration (Cmax) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Time to Maximum Concentration (Tmax) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Area Under the Concentration-Time Curve From Time Zero to the End of the Dosing Interval (AUClast) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Area Under the Concentration-Time Curve From Time Zero to the End of the Dosing Interval (AUCtau) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Area Under the Concentration-Time Curve From Time Zero to Infinity (AUCinf) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Apparent Terminal Elimination Half-Life (Thalf) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Apparent Clearance (CL) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Apparent Volume of Distribution (Vss) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Accumulation Index (AI) of ADCT-901 Total Antibody, Pyrrolobenzodiazepine (PBD)-Conjugated Antibody, and Unconjugated Warhead SG3199 in Serum | Up to approximately 2.5 years
Number of Participants with an Anti-drug Antibody (ADA) Response to ADCT-901 | Up to approximately 2.5 years

CONTACTS AND LOCATIONS:
Locations (13):
- United States (7):
  - Sarah Cannon at HealthONE, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University Hospitals of Cleveland Medical Center (UHCMC), Cleveland, Ohio
  - Sarah Cannon at University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - NEXT Oncology, San Antonio, Texas
- Spain (4):
  - Institut Catala D'oncologia (ICO) - Hospital Duran I Reynals Location, Badalona, Barcelona
  - Hospital Universitari Vall D'hebron - Vall D'hebron Institut D'oncologia (VHIO), Barcelona
  - (START) Madrid - Hospital Universitario Fundación Jiménez Díaz Location, Madrid
  - Universidad Complutense de Madrid - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust - St Mary's Hospital, London, England
  - Sarah Cannon Research Institute (SCRI) - London (SCRI-UK), London, England

IPD SHARING:
Plan to Share IPD: No